CLINICAL TRIAL: NCT07243925
Title: Effect of Family Involvement Intervention on Anxiety, Independence, and Psychological Resilience in CABG Surgery Patients
Acronym: CABG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ozkan Sir, PhD, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CABG-FAMINT-TR-2025
Record Dates: First submitted 2025-09-22; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Family Size; Coronary Artery Disease
Keywords: family; coronary; family involvement
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Involvement Intervention Group (Experimental): Family Involvement Intervention Group
  Interventions: Other: Family Involvement-Based Nursing Intervention
- Standard Care Control Group (No Intervention): Standard Care Control Group

INTERVENTIONS:
Other: Family Involvement-Based Nursing Intervention — The intervention process began with the identification of a family member who could actively participate in the patient's care. These individuals were typically defined as spouses, children, siblings, or close relatives living together. Patients included in the study were admitted to the cardiovascular surgery ward approximately three days before the planned surgery. During this period, routine preoperative preparations were carried out for the patients. These preparations included carotid and saphenous vein Doppler ultrasonography, consultations with the pulmonary medicine and cardiology departments, and preoperative blood preparation
  Other Names: Family Group
  Arms: Family Involvement Intervention Group

SUMMARY:
This randomized controlled trial was conducted to examine the effect of a family-based intervention prior to coronary artery bypass grafting (CABG) surgery on patients' psychosocial and functional outcomes. In the intervention group, family members who would participate in the care process received structured training, and their active participation in the pre- and post-operative care process was ensured. The control group received standard care.

The study found that the family-based intervention reduced patients' preoperative anxiety levels, supported their independence, and strengthened their psychological resilience. The findings suggest that encouraging family involvement in patient care prior to CABG surgery can significantly contribute to both improving psychosocial adjustment and supporting the recovery process.

DETAILED DESCRIPTION:
Coronary Artery Bypass Grafting (CABG) surgery is a life-saving intervention in the treatment of cardiac diseases; however, it poses significant psychosocial and functional challenges for patients. In the preoperative period, uncertainty, fear of death, and concerns regarding recovery increase patients' anxiety levels, while in the postoperative period, loss of independence, limitations in daily living activities, and decreased psychological resilience are frequently observed. Existing literature predominantly focuses on pharmacological approaches or standard care practices for managing these issues, while studies systematically examining family involvement as an intervention model remain limited. This study evaluated the effects of a family involvement-based structured intervention on anxiety, independence, and psychological resilience in patients undergoing CABG surgery, using a randomized controlled design. Within the intervention, first-degree family members who would participate in the patient's care received training covering the surgical process, care needs, and psychosocial support strategies, and were actively engaged in both pre- and postoperative patient care. The results demonstrated that the family involvement-based intervention significantly reduced patients' anxiety, enhanced independence, and improved psychological resilience. These findings highlight that family involvement contributes not only to the physical care of CABG patients but also to their psychosocial adaptation and recovery processes. As one of the first studies to address these dimensions simultaneously, this research provides an original contribution to strengthening family-centered care in nursing practice and restructuring surgical patient care protocols.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Undergoing CABG surgery for the first time
* Being conscious and able to communicate
* Voluntarily agreeing to participate
* Having at least one family member who is able to be involved in the patient care process

Exclusion Criteria:

* Having a severe cognitive or psychiatric disorder
* Requiring prolonged intensive care admission due to postoperative complications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative Anxiety Level | Measured on the day before surgery
  Patients' anxiety levels prior to coronary artery bypass graft (CABG) surgery will be assessed using the State Anxiety Scale (SAS). The scale consists of 20 items and yields scores ranging from 20 to 80; higher scores indicate higher anxiety levels. The measurement will be conducted in person 24 hours before the surgical procedure.
Psychological Resilience Assessed by the Brief Resilience Scale (BRS) | The day before the surgery
  Participants' psychological resilience levels will be assessed using the Brief Resilience Scale (BRS). The scale consists of 6 items and is scored on a 1-5 point scale. The average score is calculated; higher scores indicate stronger psychological resilience. The measurement will be taken prior to the surgical procedure (24 hours beforehand).

SECONDARY OUTCOMES:
Functional Independence in Activities of Daily Living Assessed by the Modified Barthel Index (MBI) | The measurement is taken upon discharge from the hospital (approximately 5-7 days after surgery).
  Participants' levels of independence in daily living activities will be assessed using the Modified Barthel Index (MBI). The MBI measures 10 basic activities of daily living (e.g., eating, bathing, dressing, mobility, toileting). The score range is 0-100; a higher score indicates greater independence. The measurement is taken upon discharge from the hospital (approximately 5-7 days after surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- VAN, Erzurum, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, IPD will not be shared